CLINICAL TRIAL: NCT03451877
Title: TGFB1 and LAMA1 Gene Polymorphisms in Turkish Children With High Myopia
Brief Title: TGFB1 And LAMA1 Gene Polymorphisms in High Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Elif Demirkilinc Biler, Co-investigator, Ege University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: 2013-TIP-097
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: High Myopia; Gene Mutations
Keywords: High myopia; TGFB1Gene Polymorphisms; LAMA1 Gene Polymorphisms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Children with cycloplegia refractive error more than -6 D TGFB1 AND LAMA1 GENE POLYMORPHISMS were examined
  Interventions: Genetic: TGFB1 AND LAMA1 GENE POLYMORPHISMS
- Control group (Other): Emmetropic children TGFB1 AND LAMA1 GENE POLYMORPHISMS were examined
  Interventions: Genetic: TGFB1 AND LAMA1 GENE POLYMORPHISMS

INTERVENTIONS:
Genetic: TGFB1 AND LAMA1 GENE POLYMORPHISMS — we evaluated polymorphisms in the LAMA1 (rs2089760) and TGFB1 (rs4803455) genes in children younger than 13 years of age with ≥6 D myopia in an attempt to further elucidate the genetic basis of high myopia.

SUMMARY:
The investigators aimed to investigate TGFB1 and LAMA1 gene polymorphisms in children with high myopia in order to determine the genetic basis of large myopic shifts causing severe visual impairment and complications.

Seventy-four children with high myopia (≥6 diopters [D]; study group) and 77 emmetropic children (±0.5D; control group) were included. Genetic and polymorphism analyses were performed in the Medical Genetics Laboratory using DNA purified from the patients' blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the age of 13
* Patients with cycloplegic refraction values ≥6 D (for study group)
* Emmetropic patients (for control group)

Exclusion Criteria:

* Patients who had additional ocular pathology that may affect refraction (such as glaucoma, cataracts, corneal disease)
* Patients with history of ocular surgery

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Genetic basis of high myopia | 4 years
  evaluated polymorphisms in the LAMA1 (rs2089760) and TGFB1 (rs4803455) genes in children younger than 13 years of age with ≥6 D myopia

IPD SHARING:
Plan to Share IPD: No